CLINICAL TRIAL: NCT01539317
Title: Therapy to Prevent Sexual Pain in Menopausal Survivors of Breast Cancer
Brief Title: Therapy to Prevent Sexual Pain in Breast Cancer Survivors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Martha Goetsch, Assistant Professor, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OHSU IRB 7630
Record Dates: First submitted 2011-12-21; First posted 2012-02-27 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Vulvodynia; Dyspareunia; Breast Cancer; Menopause
Keywords: Vulvodynia; Dyspareunia; Breast Cancer; Menopause; Vaginal dryness; Painful intercourse
MeSH Terms: conditions — Vulvodynia; Dyspareunia; Breast Neoplasms | interventions — Sodium Chloride; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical liquid lidocaine (Active Comparator)
  Interventions: Drug: Topical liquid lidocaine; Drug: Topical saline
- Topical Saline (Placebo Comparator)
  Interventions: Drug: Topical liquid lidocaine; Drug: Topical saline

INTERVENTIONS:
Drug: Topical liquid lidocaine — active intervention drug numbs the hypersensitive mucosa of the vulvar vestibule
Drug: Topical saline — saline applied to the vestibule mucosa will not reverse the local tenderness
  Other Names: water

SUMMARY:
The purpose of this protocol is to determine whether pain with sexual intercourse can be reduced in menopausal, breast cancer survivors and to evaluate the effectiveness of a non-hormonal therapy (Lidocaine Liquid) vs. a placebo liquid in reducing pain.

The investigators hypothesize that the pain arises in the vulvar vestibule. The investigators predict that the localized use of lidocaine will be more efficacious than use of placebo liquid.

DETAILED DESCRIPTION:
For this study there will be three visits over a 3 month period. Subjects will undergo a gynecological exam at the screening visit to determine the severity of pain associated with uncomfortable intercourse. A touch test using Q-tips will be used during screening exam so subjects can report pain during application of both study drug and placebo. Subjects will also report pain during tampon test. A sample of vaginal cells and liquid will be obtained at screening visit so that PI can rule out possible infection, disease, or disorders. PI will also show subject the area of the vestibule in a mirror so that subject can apply study drug at home properly. Subjects will fill out 4 questionnaires about medical and health history, cancer history, pain, and distress and sexual activity. Subject will be given a supply of either study drug or placebo to take home. The first visit will last approximately 2 hours.

Subjects will return for a second visit after 4 weeks and a third visit after 8 weeks for diary review, questionnaires, and examination. The second and third visit examinations will be repeats of the examination done at the first visit, but there will be no comparison with placebo, the PI will use only study drug during the touch test. The second and third visits will last approximately 1 hour.

Subjects will fill out questionnaires throughout study participation. Topics include; medical and health history, cancer history, pain, distress and sexual activity. Subjects will also fill out a diary that charts tampon test completed from home, sexual activity performed, pain levels and study drug application days.

ELIGIBILITY:
Eligibility Criteria

1. Women aged 18 to 70 years old.
2. Has a previous diagnosis of breast cancer (ductal or lobular carcinoma, invasive).
3. 1 year from diagnosis of breast cancer.
4. Stable heterosexual partnership =/>5 years or by investigator discretion.
5. More than 6 months of consistent insertional pain with intercourse (may have stopped having intercourse due to this consistent experience of pain).
6. Menopausal, demonstrated by at least one of the following:

   i. cessation of menses for 1 years ii. Bilateral oophorectomy iii. Follicle Stimulating Hormone (FSH) level >25 in women below age 50 with an ovary and scarred or absent uterus (acceptable FSH levels can be inferred if the woman's oncologist monitors FSH during aromatase inhibitor therapy).
7. Willingness to enter a study comparing a topical placebo liquid to topical liquid lidocaine.
8. Willingness to evaluate the liquids by use of a tampon test as many as 4 times per month, and willingness to attempt intercourse if the tampon test indicates tolerable penetrative pain.

3.2 Exclusion Criteria

1. Diagnosis of benign or malignant phyllodes tumor of the breast.
2. Consistently has pain in the pelvis or low abdomen during or after intercourse (deep dyspareunia).
3. Has developed shrinkage of the vaginal opening or vaginal length to the point of being too small to succeed in having vaginal penetration with the partner (will also be assessed at the clinical exam).
4. Partner has a problem of sexual dysfunction limiting his performance or making it inconsistent.
5. The potential subject or her partner has a serious current medical condition that might interrupt completion of a 6 month study.
6. Potential subject has been diagnosed by a physical therapist with significant pelvic floor muscle dysfunction causing pain (pelvic floor myalgia).
7. Potential subject has used topical or systemic estrogen within the last 4 months.
8. Has continued tenderness of vestibule mucosa immediately after application of both test liquids.
9. Allergy to lidocaine or other numbing agents.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Goetsch, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Goetsch MF, Lim JY, Caughey AB. A Practical Solution for Dyspareunia in Breast Cancer Survivors: A Randomized Controlled Trial. J Clin Oncol. 2015 Oct 20;33(30):3394-400. doi: 10.1200/JCO.2014.60.7366. Epub 2015 Jul 27. PMID 26215946
- [Derived] Goetsch MF, Lim JY, Caughey AB. Locating pain in breast cancer survivors experiencing dyspareunia: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1231-1236. doi: 10.1097/AOG.0000000000000283. PMID 24807329
- See also: Related Info — http://www.ohsu.edu/xd/health/services/women/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2012 to June 2013; Women's Health Research Unit (WHRU) at Oregon Health and Science University (OHSU) in Portland, OR
Groups:
- Topical Liquid Lidocaine; Topical Saline: Topical liquid lidocaine: Comparison of topical liquid lidocaine to placebo on application to the vulvar vestibule
Period: Overall Study
Arm/Group | Topical Liquid Lidocaine | Topical Saline
Started | 25 | 25
Completed | 24 | 25
Not Completed | 1 | 0
Not completed — Screening Error. Deleted from analysis. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Liquid Lidocaine | Topical Saline | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.5) | 54.7 (8.9) | 55.34 (8.77)
Sex/Gender, Customized [Number; unit: participants]
  Female | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 22 | 22 | 44
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Entry Dyspareunia With Non-hormonal Therapy
Description: Mean intercourse pain reported by subjects using the Numerical Rating Scale pain ratings (range 0-10, 0 being "no pain" and 10 being "worst possible pain"). Testing was during weeks 0-4 (Phase II) (with blinded randomization for placebo vs active intervention medication) and testing was during weeks 5-12 (Phase III) (with open-label active medication for 8 weeks after completing the blinded 4 weeks). Subjects agreed to try penetration twice per week and score their pain using the Numerical Rating Scale pain ratings.The scores were averaged during each phase.
Time Frame: During Phase II (0-4 weeks) and during Phase III (5-12 weeks)
Measure: Mean (Inter-Quartile Range); unit: Units on a scale
Groups:
- Open Label: During Open-label Lidocaine 8 weeks
  Each prior arm converted to use of open label lidocaine for 2 further months.
Arm/Group | Topical Saline | Topical Liquid Lidocaine | Open Label
Number analyzed (Participants) | 21 | 22 | 41
Units on a scale
  Phase II | 5.3 [3 to 7] | 1.04 [0.65 to 1.92] | NA [NA to NA] — Phase II was not the open label portion of the study
  Phase III | 0.57 [0.07 to 1.80] | 0.45 [0 to 1.14] | 0.48 [0 to 1.78]
Statistical Analysis 1: Comparison: Topical Saline vs Topical Liquid Lidocaine; Phase II: During Blinded 4 weeks; Test type: Superiority or Other; p = 0.0149, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Topical Saline vs Topical Liquid Lidocaine vs Open Label; Phase III; Test type: Superiority or Other; p = 0.412, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Improvement of Quality of Sexual Life - Visit 1
Description: To determine whether women's quality of sexual life is improved by use of this local therapy to prevent pain with intercourse. Measured by average scores on the Sexual Function Questionnaire. There are 8 domains measured in the Sexual Function Questionnaire each asking for a score for the prior 30 days: Desire (score range 5-31; ≥23 considered normal function), Arousal-sensation (score range 4-20; ≥14 considered normal function), Arousal-lubrication (score ranges 2-10; ≥8 considered normal function), Arousal-cognitive (score range 2-10; ≥8 considered normal function), Orgasm (score range 1-15; ≥12 considered normal function), Pain (2-15; ≥12 considered normal function), Enjoyment (score range 6-30; ≥23 considered normal function) and Partner (score range 2-10; ≥8 considered normal function).
Time Frame: Visit 1 (Enrollment)
Population: Averaged scores of Sexual Function Questionnaire Visit 1 each time scoring from the prior 30 days.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Topical Saline | Topical Liquid Lidocaine
Number analyzed (Participants) | 21 | 22
units on a scale
  Desire | 11.91 [9 to 14] | 13.87 [12 to 16]
  Arousal Sensation | 8.44 [6 to 11] | 9.15 [8 to 10]
  Arousal Lubrication | 3.92 [2 to 4] | 2.97 [2 to 4]
  Arousal Cognitive | 4.28 [4 to 5] | 4.82 [4 to 6]
  Orgasm | 5.70 [1 to 10] | 7.62 [1 to 13]
  Pain | 6.04 [4.48 to 8] | 6.29 [5 to 8.48]
  Enjoyment | 15.30 [12 to 17.68] | 17.01 [14 to 18.97]
  Partner | 7.78 [6 to 9] | 8.13 [7 to 10]
Statistical Analysis 1: Comparison: Topical Saline vs Topical Liquid Lidocaine; Desire; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Topical Saline vs Topical Liquid Lidocaine; Arousal (S); Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Topical Saline vs Topical Liquid Lidocaine; Arousal (L); Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Topical Saline vs Topical Liquid Lidocaine; Arousal (C); Test type: Superiority or Other; p = 0.28, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Topical Saline vs Topical Liquid Lidocaine; Orgasm; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Topical Saline vs Topical Liquid Lidocaine; Pain; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Topical Saline vs Topical Liquid Lidocaine; Enjoyment; Test type: Superiority or Other; p = 0.54, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Topical Saline vs Topical Liquid Lidocaine; Partner; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Location of Pain in Postmenopausal Dyspareunia
Description: To determine the specific site of vulvovaginal tenderness in menopausal breast cancer survivors who have entry dyspareunia. Examine the vulvar vestibule with a swab test to determine locations and severity of touch tenderness. Eight sites were evaluated around the vaginal opening and there location was in reference to a clock face. Measured using the Numerical Rating Scale, a scale which measures pain from 0 to 10 with 0="no pain" and 10="the worst pain you have ever felt".
Time Frame: Enrollment visit
Measure: Median (Inter-Quartile Range); unit: units on a scale from 0 to 10
Arm/Group | Topical Saline | Topical Liquid Lidocaine
Number analyzed (Participants) | 25 | 24
units on a scale from 0 to 10
  1 o'clock | 0 [0 to 0] | 0 [0 to 0]
  11 o'clock | 0 [0 to 2] | 0 [0 to 0]
  12 o'clock | 1 [0 to 4] | 0 [0 to 0]
  3 o'clock | 3 [2 to 5] | 0 [0 to 1]
  4 o'clock | 4 [3 to 6] | 0 [0 to 1]
  8 o'clock | 4 [3 to 6] | 0 [0 to 0.5]
  9 o'clock | 5 [2 to 6] | 0 [0 to 1]
  6 o'clock | 2 [1 to 4] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Topical Saline vs Topical Liquid Lidocaine; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Each of 8 site comparisons had its own P-value and a value of <0.001 was the difference at the most tender sites

4. Secondary Outcome: Improvement of Quality of Sexual Life - Visit 2
Description: To determine whether women's quality of sexual life is improved by use of this local therapy to prevent pain with intercourse. Measured by averaged scores on the Sexual Function Questionnaire. There are 8 domains measured in the Sexual Function Questionnaire each asking for a score for the prior 30 days: Desire (score range 5-31; ≥23 considered normal function), Arousal-sensation (score range 4-20; ≥14 considered normal function), Arousal-lubrication (score ranges 2-10; ≥8 considered normal function), Arousal-cognitive (score range 2-10; ≥8 considered normal function), Orgasm (score range 1-15; ≥12 considered normal function), Pain (2-15; ≥12 considered normal function), Enjoyment (score range 6-30; ≥23 considered normal function) and Partner (score range 2-10; ≥8 considered normal function).
Time Frame: Visit 2 (Week 4)
Population: Averaged scores of Sexual Function Questionnaire at Visit 2 scoring from the prior 30 days.
Measure: Mean (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Topical Saline | Topical Liquid Lidocaine
Number analyzed (Participants) | 21 | 22
Units on a scale
  Desire | 14 [11 to 17] | 16.09 [14 to 19]
  Arousal Sensation | 8.14 [5 to 10] | 11.21 [9.71 to 13]
  Arousal Lubrication | 3.59 [2 to 4] | 4.18 [2 to 4]
  Arousal Cognitive | 4.69 [4 to 6] | 5.99 [5 to 7]
  Orgasm | 5.07 [1 to 9] | 9.05 [8 to 12]
  Pain | 7.96 [6 to 9.26] | 10.50 [9.13 to 12]
  Enjoyment | 16.9 [14 to 20.54] | 19.36 [17.07 to 22.07]
  Partner | 8.62 [8 to 10] | 8.68 [8 to 10]

5. Secondary Outcome: Improvement of Quality of Sexual Life - Visit 3
Description: as for outcome 2
Time Frame: Visit 3 (End of Study)
Population: Averaged scores of Sexual Function Questionnaire at Visit 1 scoring from the prior 30 days.
Measure: Mean (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Topical Saline | Topical Liquid Lidocaine
Number analyzed (Participants) | 21 | 22
Units on a scale
  Desire | 17.79 [15 to 21] | 18.32 [16 to 21]
  Arousal Sensation | 10.89 [8 to 13] | 13.15 [11 to 15.5]
  Arousal Lubrication | 4.79 [4 to 6] | 5.2 [4 to 6.5]
  Arousal Cognitive | 5.74 [5 to 7] | 7.05 [6 to 9]
  Orgasm | 6.95 [1 to 11] | 9.5 [7 to 13]
  Pain | 11.18 [10.35 to 12] | 11.67 [9.5 to 13.68]
  Enjoyment | 20.90 [17.44 to 24.44] | 22.51 [21.2 to 24]
  Partner | 8.95 [8 to 10] | 9.36 [9 to 10]

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Topical Liquid Lidocaine | Topical Saline
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes